CLINICAL TRIAL: NCT02750683
Title: Norepinephrine Exerts an Inotropic Effect at the Early Phase of Human Septic
Brief Title: Norepinephrine Exerts an Inotropic Effect at the Early Phase of Human Septic Shock
Status: Completed | Type: Observational
Sponsor: Hopital Antoine Beclere (Other)
Responsible Party: Principal Investigator, Hamzaoui Olfa, MD, Hopital Antoine Beclere
Other Study IDs: 2011-A-01230-41
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Septic Shock
Keywords: inotropic effect, norepinephrine, septic shock,
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Norepinephrine (NE) is a potent vasopressor used in septic shock to reverse hypotension. Early infusion of NE was associated with a favorable clinical outcome in a large cohort of patients . When administered early, NE increases cardiac output (CO) in patients with septic shock . This effect was suggested to be mainly related to an increased cardiac preload via the α-adrenergic-mediated decrease in systemic venous capacitance . Whether NE exerts a positive effect on cardiac contractility through β1-adrenergic stimulation is unclear. On the one hand, the sensitivity of β1-adrenergic receptors can be abnormally reduced in septic conditions. On the other hand, such a sepsis-induced down-regulation of β1-adrenergic receptors may occur relatively late and thus, might not be observed when NE is administered early. Our study was designed to examine the inotropic effects of NE when administered in the early phase of human septic shock

DETAILED DESCRIPTION:
It is a prospective observational study, in two 15-bed intensive care units, including adult patients with septic shock who have a mean arterial pressure (MAP) < 65 mmHg within the first three hours after the start of resuscitation. For every patient, the physician taking care of the patient should have already decided to initiate NE or to increase its dose in order to achieve a MAP value of at least 65mmHg without any other change of the associated therapy (fluid administration, ventilator settings, other drugs). The study was approved by the institutional review board of our institution (Comité de Protection des Personnes, Paris-Ile-de-France VII). Informed patient (or next-of-kin) consent was obtained from all patients.

Data collection: demographic and clinical information (origin of sepsis, major elements of the clinical history) were collected. The volume of fluids administered before inclusion, the use of mechanical ventilation and the interval time between the start of resuscitation and inclusion (T0) were also recorded.

Hemodynamic data: At T0 and at T1, defined as the time a MAP value of at least 65 mmHg was reached after initiating NE (or increasing its dose), heart rate (HR), systolic arterial pressure (SAP), diastolic arterial pressure (DAP), MAP and blood lactate concentration were collected.

Transthoracic echocardiographic data: Echocardiographic measurements were performed at T0 and T1.

Transthoracic echocardiographic (TTE) examination were performed with 3.75 MHZ probe using a CX50 Philips and a Vivid i (GE Healthcare) machine. Patients were on supine flat or lateral supine positions depending on their respiratory tolerance. A four- and five-chamber apical views were used in order to collect the following variables: left ventricular ejection fraction (LVEF) calculated by the biplane method of disks summation (modified Simpson's rule), velocity-time integral (VTI) of the sub-aortic flow, tissue Doppler imaging of tricuspid annular motion (Sa), tricuspid annular plane systolic excursion (TAPSE) measured by M-mode echocardiography, the peak early (E) and late (A) transmitral flow velocity, the mean early diastolic velocity (Ea) of the lateral mitral annulus, the ratios E/A and E/Ea and tissue Doppler imaging of mean systolic velocity of the lateral mitral annulus (Sm). All the parameters were averaged over three beats or five beats in case of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Septic shock
* Mean arterial pressure<65mmHg

Exclusion Criteria:

* Age less than 18 yeras old
* Pregnancy
* moribond patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an age of more than 18 years old, admitted to intensive care unit with septic shock and a mean arterial pressure of less than 65mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The changes in left ventricular ejection fraction | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Olfa Hamzaoui, MD, Principal Investigator — Hopital Antoine Beclere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamzaoui O, Jozwiak M, Geffriaud T, Sztrymf B, Prat D, Jacobs F, Monnet X, Trouiller P, Richard C, Teboul JL. Norepinephrine exerts an inotropic effect during the early phase of human septic shock. Br J Anaesth. 2018 Mar;120(3):517-524. doi: 10.1016/j.bja.2017.11.065. Epub 2017 Nov 21. PMID 29452808